CLINICAL TRIAL: NCT04639687
Title: Food as Medicine: Evaluating the Impact of Home-delivered Vegetables and Whole Grains on Diet of Food-insecure Families
Acronym: FAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Battery Powered (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-062
Record Dates: First submitted 2019-04-29; First posted 2020-11-20 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Food Insecurity; Nutrition Poor
Keywords: randomized intervention; home-delivery intervention; vegetables; whole grains; food insecurity; diet quality
MeSH Terms: conditions — Malnutrition | interventions — Food

STUDY DESIGN:
Intervention Model Description: Group A is randomized to intermediate intervention, and change in measured outcomes is changed to that of Group B, which is a wait-list control group. Group B gets intervention later, but data contributes to follow-up up data rather than randomized controlled trial data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental): If randomized to this group, household of child and participating caregiver receives 12 weekly deliveries of vegetables plus added whole grains, along with text messages containing links to cooking instruction videos
  Interventions: Behavioral: Food as Medicine Delivery
- Wait list control (delayed intervention) (Other): If randomized to this group, participants do not get any intervention activities for the first 12 weeks, and their outcome data at V2 contribute as controls. For ethical reasons, this low-income population ultimately gets the intervention (food)later, and data after they receive the intervention contributes to follow-up data only.
  Interventions: Behavioral: Food as Medicine Delivery

INTERVENTIONS:
Behavioral: Food as Medicine Delivery — 12 consecutive weeks of home-delivered vegetables plus whole grain foods along with weekly text containing educational video

SUMMARY:
Food insecurity predisposes to poor diet, thereby increasing risk for diet-sensitive chronic disease. This trial is to evaluate the impact of a model of weekly home-delivery of locally-grown vegetables along with selected whole grains on diet among low-income children living in a household with food insecurity. The investigators plan to enroll children (10-15 years) who will participate along with their parent/caregiver. Intervention will consist of 12 weeks of weekly delivered food plus recipes and text-messaged links to cooking instruction. Dyads will be randomized (2:1) to either immediate intervention or a wait-list control group, and diet and diet-related behaviors will be assessed in-person as well as over the telephone.

DETAILED DESCRIPTION:
Children and their families who are seen at the investigators primary care clinic will be screened for eligibility by the research team study staff, and caregiver/parents will be asked a short 2-item screener about access to food. This screener has been called the "Hunger Vital Sign". When a screen for household food security is positive, caregivers are invited to participate in this study along with their child, as a dyad.

This is a randomized clinical trial. The first activity consists of an in-person visit where child and caregiver answer survey questions related to diet (specifically regarding vegetable and whole grain purchase and consumption). Anthropometrics are measured. The child has a 24-hour diet recall that is conducted in person at this visit, and then two more times in the intervening time (approximately 2 weeks). They are randomized (2:1) at this visit to either receive 12 weeks of deliveries immediately (starting in approximately 2 weeks) or after a delay of 3 months, when they serve as the delayed-intervention control group.

Immediate intervention group receives a weekly delivery of vegetables and whole grains as well as 1-2 weekly text messages that contain education such as links to cooking tips and videos.

After 3 months, both immediate intervention and the delayed intervention groups return for a second in-person visit, and complete all of the visit activities. Delayed intervention group starts their deliveries at this point.

After 3 months, the delayed intervention group returns for a third in-person visit, though the immediate intervention participants complete their follow-up survey questions over the telephone, only.

This home delivery model, done in coordination with a community-supported has been successfully-piloted in a population of low-income dyads with a child having prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* child between 10-15 at time of enrollment whose caregiver screens as positive for food insecurity during visit to primary clinic
* child must reside in household with caregiver at least 5 out of 7 days a week
* dyad must reside in Oakland, CA (delivery range for farm)

Exclusion Criteria:

* Not able to consume wheat or other grains
* Caregiver and child must have cognitive capability to complete survey materials (exclude non-verbal autistic, developmental delay)
* Unable to communicate in either English or Spanish

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
vegetable consumption (servings/day) for child | 6 months
  24-diet diet recall (total vegetables)
whole grains consumption (ounce equivalents/day) for child | 6 months
  24-diet diet recall (total vegetables)
reported total cups of vegetables per day (for adult) | 6 months
  Fruit and Vegetable checklist

SECONDARY OUTCOMES:
food security | 3 months
  Core food security module (up to 18 questions)
food security | 6 months
  Core food security module (up to 18 questions)
Body mass Index | 6 months
  Body mass index, calculated
Liking Scale (Vegetables) | 6 months
  This scale (never tried, do not like, like a little, like a lot) has been validated in children as young as 4th grade. Responses will be dichotomized to represent "Ever tried" ('Never tried' versus all other responses) and "Like it" ('Never tried' or 'do not like' versus 'like a little' and 'like a lot')
Liking Scale (Whole grains) | 6 months
  This scale (never tried, do not like, like a little, like a lot) has been validated in children as young as 4th grade. Responses will be dichotomized to represent "Ever tried" ('Never tried' versus all other responses) and "Like it" ('Never tried' or 'do not like' versus 'like a little' and 'like a lot')

CONTACTS AND LOCATIONS:
Overall Officials: June Tester, MD, MPH, Principal Investigator — Assistant Clinical Scientist
Locations (1):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No